CLINICAL TRIAL: NCT05850559
Title: Assessment of the Diagnostic Role of Serum Insulin-like Growth Factor Binding Protein-3 as a Potential Biomarker for Colorectal Cancer (CRC) in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebat Allah Galal Eldin Mabady, resident in clinical pathology department, Assiut University
Other Study IDs: ELISA and colorectal cancer
Record Dates: First submitted 2023-04-13; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: evaluation of diagnostic importance of insulin like growth factor binding protein3 in patient with recently diagnosed as Colorectal cancer — evaluation of diagnostic importance of insulin like growth factor binding protein3 in patient with recently diagnosed as Colorectal cancer by Enzyme-linked immunosorbent assay (ELISA

SUMMARY:
1. evaluation of diagnostic importance of insulin like growth factor binding protein3 in patient with recently diagnosed as Colorectal cancer
2. correlation between the diagnostic efficacy of insulin like growth factor binding protein 3 with routine marker carcinoembryonic antigen.

DETAILED DESCRIPTION:
Colorectal Cancer is the third most common cancer diagnosed in the USA and the world's fourth most deadly cancer .the incidence and the mortality rate of colorectal cancer has decreased due to effective cancer screening measures.

Besides an ageing population and dietary habits of high-income countries, unfavourable risk factors such as obesity, lack of physical exercise, and smoking increase the risk of colorectal cancer.

The incidence of early-onset colorectal cancer diagnosed in patients under the age of 50 years- has been increasing around the world.

The insulin-like growth factor (IGF) system composed of two ligands, their receptors and regulatory proteins.

IGFBPs regulate the cell cycle, and the function of IGFBPs in transcriptional regulation, DNA damage repair and apoptosis induction suggest that they are closely associated with tumour development, progression, and therapy resistance.

Insulin-like growth factor peptides play important roles in regulating cell growth, cell differentiation, and apoptosis, and have been demonstrated to promote the development of colorectal cancer.

Researchers found that IGFBP3 has the potential to be used as early indicator for colorectal cancer diagnosis.

Moreover, IGFBP3 as a risk factor for carcinogenesis has been demonstrated in many cancers.

IGFBP3 as a tumour suppressor was reported to be down-regulated in some cancers. But some other publications showed its overexpression is associated with poor prognosis for several cancers including pancreatic endocrine neoplasms.

Meanwhile, epidemiological studies indicated that higher circulating IGFBP3 level were an increased risk of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at South Egypt Cancer institute and diagnosed Colorectal cancer patients
2. Patients not went to surgery

Exclusion Criteria:

1. patients receive any anti-cancer therapy.
2. Patients diagnosed with other concomitante cancer or chronic diseases

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A calculated minimum sample of 50 patients diagnosed with Colorectal cancer and 30 apparently healthy subject with matched age and sex as acontrol group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-05 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Diagnostic Role of Serum Insulin-like Growth Factor Binding Protein-3 as a Potential Biomarker for Colorectal Cancer (CRC) in Egypt | Baseline
  measure level of insulin like growth factor binding protein3 in serum in patients of egypt recently diagnosed as Colorectal cancer by useing ELISA

REFERENCES:
- [Background] Murphy N, Carreras-Torres R, Song M, Chan AT, Martin RM, Papadimitriou N, Dimou N, Tsilidis KK, Banbury B, Bradbury KE, Besevic J, Rinaldi S, Riboli E, Cross AJ, Travis RC, Agnoli C, Albanes D, Berndt SI, Bezieau S, Bishop DT, Brenner H, Buchanan DD, Onland-Moret NC, Burnett-Hartman A, Campbell PT, Casey G, Castellvi-Bel S, Chang-Claude J, Chirlaque MD, de la Chapelle A, English D, Figueiredo JC, Gallinger SJ, Giles GG, Gruber SB, Gsur A, Hampe J, Hampel H, Harrison TA, Hoffmeister M, Hsu L, Huang WY, Huyghe JR, Jenkins MA, Keku TO, Kuhn T, Kweon SS, Le Marchand L, Li CI, Li L, Lindblom A, Martin V, Milne RL, Moreno V, Newcomb PA, Offit K, Ogino S, Ose J, Perduca V, Phipps AI, Platz EA, Potter JD, Qu C, Rennert G, Sakoda LC, Schafmayer C, Schoen RE, Slattery ML, Tangen CM, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Visvanathan K, Vodicka P, Vodickova L, Vymetalkova V, Wang H, White E, Wolk A, Woods MO, Wu AH, Zheng W, Peters U, Gunter MJ. Circulating Levels of Insulin-like Growth Factor 1 and Insulin-like Growth Factor Binding Protein 3 Associate With Risk of Colorectal Cancer Based on Serologic and Mendelian Randomization Analyses. Gastroenterology. 2020 Apr;158(5):1300-1312.e20. doi: 10.1053/j.gastro.2019.12.020. Epub 2019 Dec 27. PMID 31884074
- [Background] Pankaj J, Kumari JR, Kim W, Lee SA. Insulin-like Growth Factor-1, IGF-binding Protein-3, C-peptide and Colorectal Cancer: a Case-control Study. Asian Pac J Cancer Prev. 2015;16(9):3735-40. doi: 10.7314/apjcp.2015.16.9.3735. PMID 25987030
- [Background] Naguib R, Abouegylah M, Sharkawy S, Fayed AA, Naguib H. Evaluation of Serum Levels of Insulin-Like Growth Factor 1 and Insulin-Like Growth Factor-Binding Protein 3 in Patients With Colorectal Cancer: A Case-Control Study. Cureus. 2021 Nov 25;13(11):e19881. doi: 10.7759/cureus.19881. eCollection 2021 Nov. PMID 34858769